CLINICAL TRIAL: NCT05435963
Title: Effect of Pulmonary Rehabilitation on Reducing Loneliness in Individuals With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Impact of Pulmonary Rehabilitation on Loneliness in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AlsubheenS
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Loneliness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COPD undergoing pulmonary rehabilitation (Experimental): 45 individuals with COPD will complete the UCLA-LS scale, CRQ, HADS, and 6 minute walk test before and after pulmonary rehabilitation.
  Interventions: Behavioral: Pulmonary rehabilitation (PR)

INTERVENTIONS:
Behavioral: Pulmonary rehabilitation (PR) — A typical PR program will include exercise training, disease-specific and self-management strategies education, and will last 6 - 8 weeks

SUMMARY:
Loneliness is the feeling of sadness because one wants friends or company. This feeling is common in patients with chronic lung disease, who suffer from breathing difficulty, chronic cough, and reduced physical and mental health. These problems lead to a reduced ability for doing daily activities and cause a loss of social life. Pulmonary rehabilitation (PR) includes exercise and education. PR has been shown to improve health status in patients with chronic lung disease but its impact on loneliness levels has never been assessed. This study aims to assess the effect of PR on reducing loneliness in patients with chronic lung disease.

DETAILED DESCRIPTION:
Pulmonary rehabilitation (PR), composed of exercise training, education, and self-management strategies, is the standard of care for managing individuals with chronic obstructive pulmonary disease (COPD). PR improves dyspnea, functional exercise capacity, health-related quality of life and decreases hospitalizations and mortality. Regular exercise has been shown to reduce loneliness in older adults and those with chronic conditions, in association with a reduction in pain, the development of friendly relationships and enhanced psychological well-being. However, there is limited information regarding the impact of PR on the level of loneliness in individuals with COPD.

Study Purpose The purpose of this study is to examine the effect of PR on loneliness levels in individuals with COPD and to examine the relationship between changes in loneliness and changes in exercise capacity, health-related quality of life, depression, and anxiety levels.

This pre-post interventional study will be conducted at the West Park Healthcare Centre and St. Joseph's Healthcare Hamilton. Ethics approval will be obtained from the Joint West Park Healthcare Centre - The Salvation Army Toronto Grace Health Centre Research Ethics Board (JREB) and the Hamilton Integrated Research Ethics Board (HiREB).

Participants Based on Mimi et al. (2014), a sample size of 45 participants is required to detect minimal significant effects on the University of California & Los-Angeles Loneliness scale (UCLA-LS), with 80% power (α= 0.05, β= 0.20) and assuming a drop-out rate of 25%. The sample will include male and female individuals who have been diagnosed with COPD.

ELIGIBILITY:
Inclusion Criteria:

* A spirometry (FEV1/FVC < 0.70) or physician-confirmed diagnosis of COPD
* Aged 18 years or more
* Ability to complete at least 60% of the PR program that includes exercise, education, and behaviour change intervention
* Ability to provide written informed consent.

Abbreviations:

FEV1: forced expiratory volume in 1 second FVC: forced vital capacity

Exclusion Criteria:

* Do not have sufficient language skills (non-English speaking or reduced cognition)
* Are unable to complete at least 60% of PR
* Fail to complete the primary outcome measure, the University of California, and Los Angeles Loneliness scale (UCLA-LS).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
The University of California and Los Angeles Loneliness scale (UCLA-LS) | 10 months
  Loneliness questionnaire. The UCLA-LS is a 20-item scale used to assess loneliness in the general population. Participants respond to each item on a 1-4 Likert scale, from "never" to "always". Positively worded items are reverse scored. The scale has a possible total score of 20 to 80 points, with a higher score indicating greater loneliness

SECONDARY OUTCOMES:
Chronic Respiratory Disease Questionnaire (CRQ) | 10 months
  Quality of life questionnaire: composed of 20 items that measure the quality of life of individuals with COPD across four domains including dyspnea (five items), fatigue (four items), emotional function (seven items), and mastery (four items). Scoring for each item ranges from one (maximum impairment) to seven (no impairment), with high scores indicating less impairments.
Generalized Anxiety Disorder - 7 (GAD - 7) Measure | 10 months
  Anxiety will be assessed using the GAD - 7. The GAD - 7 is a 7 - item self-report questionnaire measuring symptoms of anxiety experienced in the preceding two weeks. Responses are assigned a score of 0, 1, 2, or 3 to reflect "not at all", "several days", "more than half the days", or "nearly everyday" respectively. A total score is calculated with scores of 5, 10 and 15 indicating mild, moderate and severe anxiety respectively.
6-Minute Walk Test | 10 months
  Measure of exercise tolerance
Patient Health Questionnaire - 9 (PHQ - 9) | 10 months
  Depression will be assessed using the PHQ - 9 23. The PHQ-9 is a 9-item self-report questionnaire measuring symptoms of depression experienced in the preceding two weeks. Responses are assigned a score of 0, 1, 2, or 3 to reflect "not at all", "several days", "more than half the days", or "nearly everyday" respectively 23. A total score is calculated with scores of 5, 10, 15 and 20 indicating mild, moderate, moderately severe and severe depression respectively

CONTACTS AND LOCATIONS:
Overall Officials: Dina Brooks, PhD, Principal Investigator — McMaster University
Locations (1):
- West Park Healthcare Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No